CLINICAL TRIAL: NCT03149484
Title: Remote Microphone Technology in Pediatric Bone Anchored Implant Recipients
Brief Title: Use of RM Technology in Pediatric BAI Recipients
Status: Completed | Type: Observational
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Hillary A Snapp, Assistant Professor, University of Miami
Other Study IDs: 20170224
Record Dates: First submitted 2017-05-04; First posted 2017-05-11 (Actual); Last update posted 2023-04-27 (Actual); Status verified 2023-04

CONDITIONS: Hearing Loss, Unilateral
MeSH Terms: conditions — Hearing Loss, Unilateral | interventions — Drug Delivery Systems

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (2):
- Pediatric Group: Children with unilateral conductive hearing loss who are treated with bone conductive devices
  Interventions: Device: Personal remote microphone (RM) system; Other: Subjective Questionnaire
- Parent/Guardian Group: The parent or guardian of a child with unilateral conductive hearing loss who are treated with bone conductive devices
  Interventions: Other: Subjective Questionnaire

INTERVENTIONS:
Device: Personal remote microphone (RM) system — Speech perception in noise performance will be evaluated in the unaided, bone conduction device (BAHA) aided, and bone conduction device (BAHA) + RM conditions. All test measures are non-experimental and commercially available.
  Groups: Pediatric Group
Other: Subjective Questionnaire — These subjective questionnaires will be given pre- and post-evaluation to both the subject and their guardian in order to determine the impact of RM on subject and guardian perceptions of listening in noise.

SUMMARY:
The purpose of this research study is to learn about the hearing outcomes of children with conductive hearing loss who are treated with bone conductive devices and their outcomes with remote microphone technology.

DETAILED DESCRIPTION:
The purpose of this research study is to learn about the hearing outcomes of children with unilateral conductive hearing loss who are treated with bone conductive devices and their outcomes with remote microphone technology. It has been shown that the use of intervention (hearing aids, cochlear implants, bone conduction devices) alone does not alleviate the difficulties children with hearing loss encounter in noisy environments such as a classroom or restaurant. One of the most common methods to help children hear better in these types of environments is the use of a personal remote microphone (RM) system. This study will evaluate how much benefit children are getting from their bone conduction device alone compared to the bone conduction device with a personal RM system.

ELIGIBILITY:
Inclusion Criteria:

* English speaking
* unilateral conductive hearing loss with a minimum of a 30 dB air-bone gap and their parent/guardian

Exclusion Criteria:

* Do not meet inclusion criteria

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: English speaking pediatric conduction device users ages 5 to 18 and their parent/guardian will be included for study. These pediatric patients have a unilateral conductive hearing loss with a minimum of a 30 dB air-bone gap.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2017-05-02 (Actual); Primary Completion 2019-04-11 (Actual); Study Completion 2019-04-11 (Actual)

PRIMARY OUTCOMES:
Speech Understanding in Noise | 40 minutes
  Investigate benefit of remote microphone (RM) for listening in noise in children with bone conduction hearing devices by calculating SNR loss
Parent and Child Perception of Hearing Loss Questionnaire | 20 minutes
  Determine the parent and child perception of the hearing loss and its impact pre- and post-evaluation using a subjective questionnaire created to further understand the child and parent's perception of their disability.

CONTACTS AND LOCATIONS:
Overall Officials: Hillary Snapp, AuD, Principal Investigator — University of Miami
Locations (1):
- University of Miami Department of Otolaryngology, Miami, Florida, United States